CLINICAL TRIAL: NCT06296745
Title: An Open-label, Single-arm, Phase II Trial of Intrathecal Pemetrexed for Leptomeningeal Metastasis From Lung Adenocarcinoma That Progressed After a Double Dose of Third-generation TKIs, Including Osimertinib
Brief Title: Intrathecal Pemetrexed for Leptomeningeal Metastasis From Lung Adenocarcinoma That Progressed After Osimertinib.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-008-01
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Leptomeningeal Metastasis
Keywords: Leptomeningeal metastasis; Intrathecal chemotherapy; Pemetrexed; Osimertinib; Epidermal growth factor receptor mutation; Non-small-cell lung cancer
MeSH Terms: conditions — Meningeal Carcinomatosis; Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group (Experimental): Intra-pemetrexed
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 15 mg was administered with dexamethasone 5 mg via intraventricular or via lumbar puncture. First, induction intrathecal chemotherapy, twice per week for 2 weeks; then consolidation intrathecal chemotherapy, once per week for 4 weeks; and maintenance intrathecal chemotherapy, once per month until disease progression or unmanageable drug-related toxicity.

SUMMARY:
Pemetrexed is one of the first-line chemotherapeutic agents for non-squamous non-small cell lung cancer (NSCLC). Since 2017, intrathecal pemetrexed has shown good efficacy for patients with leptomeningeal metastases from NSCLC. It has been recommended as the preferred drug for intrathecal chemotherapy by the Chinese Society of Clinical Oncology (CSCO) guidelines. Tyrosine kinase inhibitors (TKIs) play a promising role in treating non-small cell lung cancer patients with epidermal growth factor receptor (EGFR) mutations. An international multi-center clinical study published in 2019 confirmed that double dose of osimertinib showed significant improvement in leptomeningeal metastases from NSCLC with EGFR exon 19 deletion or exon 21 L858R/T790M mutation. It makes TKIs the mainstay of treatment for patients with EGFR-mutant NSCLC with leptomeningeal metastases. However, the choice of treatment after resistance to targeted therapy is a hot topic in clinical practice, with 78% of patients in the study above who responded to double-dose osimertinib still showing progression at the time of follow-up. The purpose of this study was to observe the safety and efficacy of intrathecal pemetrexed for leptomeningeal metastasis from lung adenocarcinoma that progressed after a double dose of a third-generation TKI such as osimertinib.

DETAILED DESCRIPTION:
This study is a single arm, open and phase II clinical trial. Consecutive patients with leptomeningeal metastases from lung adenocarcinoma that progressed after a double dose of a third-generation TKI such as osimertinib are enrolled in this study. Concomitant regimen consisted of intrathecal chemotherapy (via lumbar puncture, pemetrexed 15 mg, plus dexamethasone 5 mg, twice a week for 2 weeks as an induction phase, followed by once a week for 4 weeks as a consolidation phase. Thereafter, the maintenance phase is once a month). The RANO proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 75 years.
2. Histologically or cytologically confirmed diagnosis of NSCLC with single activating EGFR mutations (L858R or Exon19Del).
3. Confirmed diagnosis of leptomeningeal metastasis according to ESMO/ EANO guidelines.
4. Progression after previous double doses of third-generation TKIs such as Osimertinib.
5. Normal liver and kidney function; WBC≥4000/mm3, Plt≥100000/mm3.
6. No history of severe nervous system disease.
7. No severe dyscrasia.

Exclusion Criteria:

1. Any evidence of nervous system failure, including severe encephalopathy, grade 3 or 4 leukoencephalopathy on imaging, and Glasgow Coma Score less than 11.
2. Any evidence of extensive and lethal progressive systemic diseases without effective treatment.
3. Patients with poor compliance or other reasons that were unsuitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The response assessment in neuro-oncology criteria (RANO) proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.
Neurological progression-free survival (NPFS) | From date of treatment until the date of first documented neurological progression or date of death from any cause, whichever came first, assessed up to 6 months.
  NPFS was defined as time from the start of treatment until neurological progression or death. The neurological progression was determined based on the RANO proposal evaluation criteria which have been established and published on Neuro Oncol.

SECONDARY OUTCOMES:
Overall survival | From the enrollment of this study until date of death from any cause, whichever came first, or the last follow-up (at least 7 months).
  Survival time was recorded since the date of patient enrollment. All patients were followed up until death or the end of the study.
Incidence of treatment-related adverse events | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The incidence of treatment-related adverse events were measured for determining tolerability and safety. Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4.03). Events of grade 3-5 are defined as moderate and severe adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Pan, Principal Investigator — Guangzhou Medical University
Locations (1):
- The Affiliated Huizhou Hospital, Guangzhou Medical University, Huizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will be available to other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication.
Access Criteria: Individual participant data will be public accessable via contacting with principal investigator by email within 6 months after the trial complete.

REFERENCES:
- [Background] Yang JCH, Kim SW, Kim DW, Lee JS, Cho BC, Ahn JS, Lee DH, Kim TM, Goldman JW, Natale RB, Brown AP, Collins B, Chmielecki J, Vishwanathan K, Mendoza-Naranjo A, Ahn MJ. Osimertinib in Patients With Epidermal Growth Factor Receptor Mutation-Positive Non-Small-Cell Lung Cancer and Leptomeningeal Metastases: The BLOOM Study. J Clin Oncol. 2020 Feb 20;38(6):538-547. doi: 10.1200/JCO.19.00457. Epub 2019 Dec 6. PMID 31809241
- [Background] Pan Z, Yang G, Cui J, Li W, Li Y, Gao P, Jiang T, Sun Y, Dong L, Song Y, Zhao G. A Pilot Phase 1 Study of Intrathecal Pemetrexed for Refractory Leptomeningeal Metastases From Non-small-cell Lung Cancer. Front Oncol. 2019 Aug 30;9:838. doi: 10.3389/fonc.2019.00838. eCollection 2019. PMID 31544065
- [Background] Pan Z, Yang G, He H, Cui J, Li W, Yuan T, Chen K, Jiang T, Gao P, Sun Y, Cong X, Li Z, Wang Y, Pang X, Song Y, Zhao G. Intrathecal pemetrexed combined with involved-field radiotherapy as a first-line intra-CSF therapy for leptomeningeal metastases from solid tumors: a phase I/II study. Ther Adv Med Oncol. 2020 Jul 17;12:1758835920937953. doi: 10.1177/1758835920937953. eCollection 2020. PMID 32733606
- [Background] Xu Z, Hao X, Wang Q, Yang K, Li J, Xing P. Intracranial efficacy and safety of furmonertinib 160 mg with or without anti-angiogenic agent in advanced NSCLC patients with BM/LM as salvage therapy. BMC Cancer. 2023 Mar 4;23(1):206. doi: 10.1186/s12885-023-10676-x. PMID 36870951